CLINICAL TRIAL: NCT00642915
Title: A 24 Week, Open-Label, Single Arm, Multi-Center Clinical Study to Document the Benefits of the Combination of Lantus and Amaryl in Ethnic Japanese Type 2 Diabetic Patients Living Outside of Japan (in US or Brazil), Who Failed Good Metabolic Control With Oral Antidiabetic Drugs (OADs)
Brief Title: Insulin Glargine Benefits in Japanese Pts Outside of Japan (US or Brazil)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, Sanofi-Aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4039
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine; glimepiride

INTERVENTIONS:
Drug: Lantus, Amaryl
  Other Names: insulin glargine,glimepiride

SUMMARY:
To estimate the efficacy of combination therapy with Lantus plus Amaryl in controlling blood glucose in Japanese patients with type 2 diabetes having failed OAD therapy, and document the ability to preserve the endocrine pancreatic function with Lantus plus Amaryl combination therapy

ELIGIBILITY:
Inclusion Criteria:

* All patients planned for enrollment into this study had to have noninsulin-dependent diabetes mellitus (NIDDM) (type 2 diabetes) and were not able to maintain good metabolic control with OADs.
* Enrolled patients could be male or female, of documented Japanese ethnic origin, and between the ages of 20 and 70 years, inclusive.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-06; Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Estimate the efficacy of combination therapy with Lantus plus Amarylin controlling blood glucose in Japanese patients with type 2 diabetes having failed oral antidiabetic drug therapy | Hemoglobin A1c values were measured at Screening and at every visit thereafter.

SECONDARY OUTCOMES:
Document the ability to preserve the endocrine pancreatic function with Lantus plus Amaryl combination therapy | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tadaaki Karino, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, São Paulo, Brazil

REFERENCES:
- [Background] Kawamori R, Eliaschewitz FG, Takayama H, Hayashida CY. Efficacy of insulin glargine and glimepiride in controlling blood glucose of ethnic Japanese patients with type 2 diabetes mellitus. Diabetes Res Clin Pract. 2008 Jan;79(1):97-102. doi: 10.1016/j.diabres.2007.08.007. Epub 2007 Oct 4. PMID 17919763